CLINICAL TRIAL: NCT04921267
Title: Impacts of Training on Effortful Listening
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Kansas State University (Other)
Responsible Party: Principal Investigator, Matthew Wisniewski, Assistant Professor, Kansas State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB9406
Record Dates: First submitted 2020-03-11; First posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Training Group

STUDY DESIGN:
Intervention Model Description: 2 groups. One group is trained to listening through simulated hearing protection. The other receives no such training.
Who Masked: Participant
Masking Description: Participant doesn't know what condition they are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- trained group (Experimental): group receives training with sounds that correspond to simulated hearing protection
  Interventions: Behavioral: training
- Control (No Intervention): group receives no training

INTERVENTIONS:
Behavioral: training — training with filtered speech
  Arms: trained group

SUMMARY:
Human listeners will hear speech masked by single-talker speech before and after auditory training.

DETAILED DESCRIPTION:
Human listeners will hear speech masked by single-talker speech before and after auditory training. Training-related changes in EEG dynamics and behavioral measures of accuracy and effort will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* normal hearing

Exclusion Criteria:

* hearing loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
pretest EEG alpha power | one day before training
  power in the alpha-band
posttest EEG alpha power | one day after training
  power in the alpha-band
pretest accuracy | one day before training
  proportion correct for identifying speech
posttest accuracy | one day after training
  proportion correct for identifying speech

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Wisniewski, PhD, Principal Investigator — Kansas State University
Locations (1):
- Kansas State University, Manhattan, Kansas, United States

IPD SHARING:
Plan to Share IPD: No